CLINICAL TRIAL: NCT00996294
Title: Surgical Treatment of Type 2 Diabetes Mellitus in Patients With BMI <35 kg/m2 (Italian Title: "La Terapia Chirurgica Del Diabete Mellito di Tipo 2 Nel Paziente Con BMI Inferiore a 35 kg/m2")
Brief Title: Surgical Treatment of Type 2 Diabetes Mellitus in <35 Body Mass Index (BMI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Nicola Scopinaro, Azienda Ospedaliera Universitaria "San Martino", Genova, Italy
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIA-CHIR
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-10

CONDITIONS: Type 2 Diabetes Mellitus; Bariatric Surgery; Biliopancreatic Diversion; Gastric Bypass
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Biliopancreatic Diversion; Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgery (Experimental): patients will be submitted to biliopancreatic diversion or gastric bypass
  Interventions: Procedure: biliopancreatic diversion, gastric bypass

INTERVENTIONS:
Procedure: biliopancreatic diversion, gastric bypass — biliopancreatic diversion consists of a distal gastrectomy with a long Roux-en-Y reconstruction, where the enteroenterostomy is placed 50 cm proximal to the ileocecal valve gastric bypass consists of creating a small proximal gastric pouch by division of the upper stomach, with reconstruction of the GI continuity by means of a Roux-en-Y loop

SUMMARY:
Thirty type 2 diabetic patients will be submitted to biliopancreatic diversion and 20 to gastric bypass. Subjects will be monitored during a 5 year period to assess the effects of the operations on diabetes control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Duration of diabetes ≥ 3 years
* Poor glycemic control (i.e., HbA1c ≥ 7.5%) in spite of hypoglycemic therapy in accordance with good clinical practice (GCP)

Exclusion Criteria:

* Specific contraindication to obesity surgery or biliopancreatic diversion or gastric bypass
* Pregnancy
* Medical conditions requiring acute hospitalisation
* Severe diabetes complications or associated medical conditions [such as blindness, end-stage renal failure (i.e. serum creatinine >2 mg/dl), liver cirrhosis, malignancy, chronic congestive heart failure (NYHA class III and IV)]
* Recent (within preceding 12 months) myocardial infarction, stroke or TIA
* Unstable angina pectoris
* Psychological conditions which may hamper patient's cooperation
* Geographic inaccessibility
* Any condition which, in the judgment of the Investigator, may make risky the participation in the study or bias the results

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2009-10 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Diabetes control, define by FSG and HbA1c | 1 year

SECONDARY OUTCOMES:
Diabetes control defined by FSG and HbA1c | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Scopinaro, MD, Principal Investigator — Azienda Ospedaliera Universitaria "San Martino", Genova, Italy
Locations (1):
- Ospedale San Martino, Genova, Italy

REFERENCES:
- [Derived] Scopinaro N, Adami GF, Papadia FS, Camerini G, Carlini F, Briatore L, Andraghetti G, Catalano M, Cordera R. Effects of gastric bypass on type 2 diabetes in patients with BMI 30 to 35. Obes Surg. 2014 Jul;24(7):1036-43. doi: 10.1007/s11695-014-1206-1. PMID 24647849
- [Derived] Scopinaro N, Adami GF, Papadia FS, Camerini G, Carlini F, Briatore L, D'Alessandro G, Parodi C, Weiss A, Andraghetti G, Catalano M, Cordera R. The effects of biliopancreatic diversion on type 2 diabetes mellitus in patients with mild obesity (BMI 30-35 kg/m2) and simple overweight (BMI 25-30 kg/m2): a prospective controlled study. Obes Surg. 2011 Jul;21(7):880-8. doi: 10.1007/s11695-011-0407-0. PMID 21541815
- [Derived] Scopinaro N, Adami GF, Papadia FS, Camerini G, Carlini F, Fried M, Briatore L, D'Alessandro G, Andraghetti G, Cordera R. Effects of biliopanceratic diversion on type 2 diabetes in patients with BMI 25 to 35. Ann Surg. 2011 Apr;253(4):699-703. doi: 10.1097/SLA.0b013e318203ae44. PMID 21475009